CLINICAL TRIAL: NCT03838510
Title: Repeated-dose Behavioral Intervention to Reduce Opioid Overdose: A Two-Site Randomized-Controlled Efficacy Trial (REBOOT)
Brief Title: Repeated-dose Behavioral Intervention to Reduce Opioid Overdose
Acronym: REBOOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Francisco Department of Public Health (Other Government)
Responsible Party: Principal Investigator, Phillip Coffin, MD, MIA, Director, Substance Use Research Unit, San Francisco Department of Public Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5R01DA045690-02 (NIH)
Record Dates: First submitted 2019-02-07; First posted 2019-02-12 (Actual); Results first posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Opioid-Related Disorders; Drug Overdose
MeSH Terms: conditions — Opioid-Related Disorders; Drug Overdose

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Counseling Intervention (Experimental)
  Interventions: Behavioral: REBOOT
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: REBOOT — The brief counseling intervention will utilize Motivational Interviewing and skills-building techniques to modify personal overdose risk behaviors and develop skills as a peer responder for witnessed overdose. The counselor will draw upon themes of safer substance use to address overdose risk behaviors and determine readiness for change in substance use.
  Arms: Brief Counseling Intervention

SUMMARY:
REBOOT is a randomized trial of a repeated-dose brief intervention to reduce overdose and risk behaviors among naloxone recipients with opioid use disorder. It includes an established overdose education curriculum within an Informational-Motivation-Behavior (IMB) model. This study will test the efficacy of REBOOT vs attention-control.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Characteristics of opioid use history
* Previously received take-home naloxone
* No life-threatening illness likely to progress clinically during trial
* Able/willing to provide informed consent and locator information, communicate in English, and adhere to visit schedule

Exclusion Criteria:

* Suicidal ideation
* Participating in another interventional study that could possibly impact the study's outcomes of interest
* Planning to leave San Francisco/Boston metro area during study
* Previously exposed to REBOOT counseling intervention
* Any condition that, in the Principal Investigator's judgment, interferes with safe study participation or adherence to study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip O Coffin, MD, MIA, Principal Investigator — San Francisco Department of Public Health
Locations (2):
- United States (2):
  - San Francisco Department of Public Health, San Francisco, California
  - Boston Medical Center, Boston, Massachusetts

REFERENCES:
- [Derived] Harris MTH, Laks J, Hurstak E, Jain JP, Lambert AM, Maschke AD, Bagley SM, Farley J, Coffin PO, McMahan VM, Barrett C, Walley AY, Gunn CM. "If you're strung out and female, they will take advantage of you": A qualitative study exploring drug use and substance use service experiences among women in Boston and San Francisco. J Subst Use Addict Treat. 2024 Feb;157:209190. doi: 10.1016/j.josat.2023.209190. Epub 2023 Oct 20. PMID 37866442
- [Derived] McMahan VM, Arenander J, Matheson T, Lambert AM, Brennan S, Green TC, Walley AY, Coffin PO. "There's No Heroin Around Anymore. It's All Fentanyl." Adaptation of an Opioid Overdose Prevention Counseling Approach to Address Fentanyl Overdose: Formative Study. JMIR Form Res. 2022 Sep 7;6(9):e37483. doi: 10.2196/37483. PMID 36069781

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: The attention control group will watch a show or listen to a podcast for the same time duration as the intervention sessions.
Period: Overall Study
Arm/Group | Brief Counseling Intervention | Control Group
Started | 133 | 135
Completed | 112 | 121
Not Completed | 21 | 14

BASELINE CHARACTERISTICS:
Groups:
- Control Group: Participants in the control group will watch a show or listen to a podcast for the same amount of time as an intervention session as an attention control.
- Total: Total of all reporting groups
Arm/Group | Brief Counseling Intervention | Control Group | Total
Number analyzed (Participants) | 133 | 135 | 268
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (10.2) | 41.7 (9.9) | 43 (10)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 86 | 79 | 165
  Female | 46 | 54 | 100
  Trans female | 1 | 1 | 2
  Trans male | 0 | 0 | 0
  Other | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 22 | 39
  Not Hispanic or Latino | 116 | 110 | 226
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 6
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 19 | 37
  White | 90 | 84 | 174
  More than one race | 10 | 15 | 25
  Unknown or Not Reported | 9 | 14 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 133 | 135 | 268

OUTCOME MEASURES:

1. Primary Outcome: Number of Overdose Events
Description: Number of overdose events will be measured by self-report via timeline follow-back (TLFB) assessment, ED/EMS records, and Vital records.
Time Frame: 16 Months
Measure: Median (Inter-Quartile Range); unit: overdoses
Arm/Group | Brief Counseling Intervention | Control Group
Number analyzed (Participants) | 133 | 135
overdoses | 0 [0 to 1] | 0 [0 to 1]

ADVERSE EVENTS:
Time Frame: 16 months
Arm/Group | Brief Counseling Intervention | Control Group
All-Cause Mortality (participants affected / at risk) | 4/133 | 4/135
Serious Adverse Events (participants affected / at risk) | 88/133 | 78/135
Other Adverse Events (participants affected / at risk) | 69/133 | 60/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brief Counseling Intervention (N=133) | Control Group (N=135)
heart failure (Cardiac disorders) | 0 | 1
heart attack (Cardiac disorders) | 0 | 1
hernia (Gastrointestinal disorders) | 0 | 1
norovirus (Gastrointestinal disorders) | 0 | 1
gallstone (Hepatobiliary disorders) | 0 | 1
gallbladder infection (Hepatobiliary disorders) | 0 | 1
adverse reaction to medication (Immune system disorders) | 0 | 1
endocarditis (Infections and infestations) | 0 | 1
muscle infection (Infections and infestations) | 0 | 1
hand infection (Infections and infestations) | 0 | 1
blood infection (Infections and infestations) | 0 | 1
pneumonia (Infections and infestations) | 0 | 1
upper respiratory infection (Infections and infestations) | 0 | 1
soft tissue infection (Infections and infestations) | 0 | 1
UTI (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
abcess (Infections and infestations) | 0 | 1
excessive sweating/fever (Infections and infestations) | 0 | 1
car accident (Injury, poisoning and procedural complications) | 0 | 1
fall (Injury, poisoning and procedural complications) | 0 | 1
head injury (Injury, poisoning and procedural complications) | 0 | 1
overdose (Injury, poisoning and procedural complications) | 0 | 1
broken wrist (Injury, poisoning and procedural complications) | 0 | 1
physical assault (Injury, poisoning and procedural complications) | 0 | 1
dislocated shoulder (Injury, poisoning and procedural complications) | 0 | 1
blood poisoning and kidney failure (Injury, poisoning and procedural complications) | 0 | 1
car accident (Musculoskeletal and connective tissue disorders) | 0 | 1
broken ankle (Musculoskeletal and connective tissue disorders) | 0 | 1
back and shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 1
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
seizure (Nervous system disorders) | 0 | 1
memory loss and headache (Nervous system disorders) | 0 | 1
confusion, loss of balance, slurred speech (Nervous system disorders) | 0 | 1
coma (Nervous system disorders) | 0 | 1
suicidal ideation (Psychiatric disorders) | 0 | 1
panic attack (Psychiatric disorders) | 0 | 1
psych emergency (Psychiatric disorders) | 0 | 1
depressive episode (Psychiatric disorders) | 0 | 1
5150 hold (Psychiatric disorders) | 0 | 1
complications related to dialysis (Renal and urinary disorders) | 0 | 1
kidney failure (Renal and urinary disorders) | 0 | 1
bladder cancer (Renal and urinary disorders) | 0 | 1
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
abscess (Skin and subcutaneous tissue disorders) | 0 | 1
cellulitis (Skin and subcutaneous tissue disorders) | 0 | 1
wrist abscess (Skin and subcutaneous tissue disorders) | 0 | 1
cyst (Skin and subcutaneous tissue disorders) | 0 | 1
abscess/cellulitis (Skin and subcutaneous tissue disorders) | 0 | 1
heart murmur (Cardiac disorders) | 1 | 0
endocarditis (Cardiac disorders) | 1 | 0
overdose (Cardiac disorders) | 1 | 0
high blood sugar (Endocrine disorders) | 1 | 0
constipation (Gastrointestinal disorders) | 1 | 0
GERD (Gastrointestinal disorders) | 1 | 0
adverse reaction to medication (General disorders) | 1 | 0
sepsis (Immune system disorders) | 1 | 0
adverse reaction to medication (Immune system disorders) | 1 | 0
strep throat (Infections and infestations) | 1 | 0
tooth infection (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
fungal infection of blood (Infections and infestations) | 1 | 0
food poisoning (Infections and infestations) | 1 | 0
blood poisoning/sepsis (Infections and infestations) | 1 | 0
blood infection (Infections and infestations) | 1 | 0
soft tissue infection (Infections and infestations) | 1 | 0
knee infection (Infections and infestations) | 1 | 0
overdose (Injury, poisoning and procedural complications) | 1 | 0
car accident (Injury, poisoning and procedural complications) | 1 | 0
stabbing (Injury, poisoning and procedural complications) | 1 | 0
coma (Injury, poisoning and procedural complications) | 1 | 0
staph infection (Injury, poisoning and procedural complications) | 1 | 0
brain bruise (Injury, poisoning and procedural complications) | 1 | 0
withdrawal symptoms (Injury, poisoning and procedural complications) | 1 | 0
stimulant overdose (Injury, poisoning and procedural complications) | 1 | 0
death, suspected overdose (Injury, poisoning and procedural complications) | 1 | 0
adverse reaction to medication (Injury, poisoning and procedural complications) | 1 | 0
hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
back and hip pain (Musculoskeletal and connective tissue disorders) | 1 | 0
foot pain and swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
hip pain (Musculoskeletal and connective tissue disorders) | 1 | 0
physical assault (Musculoskeletal and connective tissue disorders) | 1 | 0
staph infection, rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
spinal fractures (Musculoskeletal and connective tissue disorders) | 1 | 0
hernia (Musculoskeletal and connective tissue disorders) | 1 | 0
head injury (Nervous system disorders) | 1 | 0
confusion/disorientation (Nervous system disorders) | 1 | 0
seizure (Nervous system disorders) | 1 | 0
stroke (Nervous system disorders) | 1 | 0
loss of consciousness (Nervous system disorders) | 1 | 0
high risk pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
mental health crisis (Psychiatric disorders) | 1 | 0
psych emergency (Psychiatric disorders) | 1 | 0
inpatient psych hold (Psychiatric disorders) | 1 | 0
kidney stone (Renal and urinary disorders) | 1 | 0
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
low oxygen (Respiratory, thoracic and mediastinal disorders) | 1 | 0
chest pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0
abscess (Skin and subcutaneous tissue disorders) | 1 | 0
staph infection (Skin and subcutaneous tissue disorders) | 1 | 0
leg infection (Skin and subcutaneous tissue disorders) | 1 | 0
foot infection (Skin and subcutaneous tissue disorders) | 1 | 0
abscess/cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0
thigh abscess (Skin and subcutaneous tissue disorders) | 1 | 0
neck abscess (Skin and subcutaneous tissue disorders) | 1 | 0
sepsis/cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0
thumb blister (Skin and subcutaneous tissue disorders) | 1 | 0
arm infection (Skin and subcutaneous tissue disorders) | 1 | 0
hysterectomy (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brief Counseling Intervention (N=133) | Control Group (N=135)
leg swelling (Blood and lymphatic system disorders) | 0 | 1
dizziness (Cardiac disorders) | 0 | 1
heart murmur (Cardiac disorders) | 0 | 1
ulcers (Gastrointestinal disorders) | 0 | 1
GI lesions/ulcers (Gastrointestinal disorders) | 0 | 1
ulcerative colitis (Gastrointestinal disorders) | 0 | 1
fatigue (General disorders) | 0 | 1
Hepatitis C infection (Infections and infestations) | 0 | 1
spinal infection (Infections and infestations) | 0 | 1
UTI (Infections and infestations) | 0 | 1
flu (Infections and infestations) | 0 | 1
toe infection (Infections and infestations) | 0 | 1
stomach flu (Infections and infestations) | 0 | 1
testicle infection (Infections and infestations) | 0 | 1
infection (Infections and infestations) | 0 | 1
knee injury (Injury, poisoning and procedural complications) | 0 | 1
back injury (Injury, poisoning and procedural complications) | 0 | 1
shoulder injury (Injury, poisoning and procedural complications) | 0 | 1
head injury (Injury, poisoning and procedural complications) | 0 | 1
broken wrist (Injury, poisoning and procedural complications) | 0 | 1
blood clots (Injury, poisoning and procedural complications) | 0 | 1
fall (Injury, poisoning and procedural complications) | 0 | 1
broken thumb (Injury, poisoning and procedural complications) | 0 | 1
physical assault (Injury, poisoning and procedural complications) | 0 | 1
dislocated shoulder (Injury, poisoning and procedural complications) | 0 | 1
unintentional weight loss (Metabolism and nutrition disorders) | 0 | 1
scoliosis worsening (Musculoskeletal and connective tissue disorders) | 0 | 1
leg pain (Musculoskeletal and connective tissue disorders) | 0 | 1
painful sciatic nerve (Musculoskeletal and connective tissue disorders) | 0 | 1
knee pain (Musculoskeletal and connective tissue disorders) | 0 | 1
arthritis in feet (Musculoskeletal and connective tissue disorders) | 0 | 1
osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
broken finger (Musculoskeletal and connective tissue disorders) | 0 | 1
losing control of hand (Nervous system disorders) | 0 | 1
pain, loss of sensation on right side of body (Nervous system disorders) | 0 | 1
neurological changes s/p stroke (Nervous system disorders) | 0 | 1
seizure (Nervous system disorders) | 0 | 1
insomnia (Psychiatric disorders) | 0 | 1
ED visit (unspecified) (Psychiatric disorders) | 0 | 1
congestion and cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
chest discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
abscess (Skin and subcutaneous tissue disorders) | 0 | 1
MRSA infection (Skin and subcutaneous tissue disorders) | 0 | 1
cellulitis (Skin and subcutaneous tissue disorders) | 0 | 1
herpes (Skin and subcutaneous tissue disorders) | 0 | 1
sublocade injection reaction (Skin and subcutaneous tissue disorders) | 0 | 1
leg wound (Skin and subcutaneous tissue disorders) | 0 | 1
psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
leg swelling (Blood and lymphatic system disorders) | 1 | 0
stomach/bowel issue (Gastrointestinal disorders) | 1 | 0
ulcerative colitis (Gastrointestinal disorders) | 1 | 0
colon pain (Gastrointestinal disorders) | 1 | 0
diarrhea (Gastrointestinal disorders) | 1 | 0
withdrawal symptoms (Gastrointestinal disorders) | 1 | 0
soreness due to dental work (General disorders) | 1 | 0
withdrawal symptoms (General disorders) | 1 | 0
allergic reaction (Immune system disorders) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
stomach virus (Infections and infestations) | 1 | 0
orchitis (Infections and infestations) | 1 | 0
chlamydia (Infections and infestations) | 1 | 0
HIV (Infections and infestations) | 1 | 0
bacterial infection (Infections and infestations) | 1 | 0
tooth pain (Infections and infestations) | 1 | 0
overdose (Injury, poisoning and procedural complications) | 1 | 0
bike accident (Injury, poisoning and procedural complications) | 1 | 0
car accident (Injury, poisoning and procedural complications) | 1 | 0
injury due to physical assault (Injury, poisoning and procedural complications) | 1 | 0
headache due to physical assault (Injury, poisoning and procedural complications) | 1 | 0
sprained ankle (Injury, poisoning and procedural complications) | 1 | 0
burn (Injury, poisoning and procedural complications) | 1 | 0
knee injury (Injury, poisoning and procedural complications) | 1 | 0
injury from fall (Injury, poisoning and procedural complications) | 1 | 0
pulled muscle (Injury, poisoning and procedural complications) | 1 | 0
lost teeth due to injury (Injury, poisoning and procedural complications) | 1 | 0
dog bite (Injury, poisoning and procedural complications) | 1 | 0
knife injury (Injury, poisoning and procedural complications) | 1 | 0
broken foot (Injury, poisoning and procedural complications) | 1 | 0
hand injury (Injury, poisoning and procedural complications) | 1 | 0
physical assault (Injury, poisoning and procedural complications) | 1 | 0
unintentional weight gain (Metabolism and nutrition disorders) | 1 | 0
unintentional weight loss (Metabolism and nutrition disorders) | 1 | 0
broken cast (Musculoskeletal and connective tissue disorders) | 1 | 0
hip pain (Musculoskeletal and connective tissue disorders) | 1 | 0
hip pain/arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
nervous twitching (Nervous system disorders) | 1 | 0
anxiety attack (Psychiatric disorders) | 1 | 0
painful menstruation (Reproductive system and breast disorders) | 1 | 0
cervical polyp (Reproductive system and breast disorders) | 1 | 0
HPV infection (Reproductive system and breast disorders) | 1 | 0
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
chest pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
lump in neck (Skin and subcutaneous tissue disorders) | 1 | 0
swollen feet (Skin and subcutaneous tissue disorders) | 1 | 0
abscess (Skin and subcutaneous tissue disorders) | 1 | 0
rash/lesions (Skin and subcutaneous tissue disorders) | 1 | 0
wound due to injection (Skin and subcutaneous tissue disorders) | 1 | 0
leg infection (Skin and subcutaneous tissue disorders) | 1 | 0
cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0
swollen eye (Skin and subcutaneous tissue disorders) | 1 | 0
infection (Skin and subcutaneous tissue disorders) | 1 | 0
blood infection/abscess (Skin and subcutaneous tissue disorders) | 1 | 0
needle stick (Social circumstances) | 1 | 0
blood clot (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT03838510/Prot_SAP_000.pdf